CLINICAL TRIAL: NCT00257114
Title: Evaluation of VELCADE (Botezomib) for Injection Employed as Re-Treatment for Efficacy, Safety, and Tolerability
Brief Title: Evaluation of VELCADE Given as Retreatment to Multiple Myeloma Patients for Efficacy, Safety and Tolerability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C05004
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Retreatment; VELCADE
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
Multiple myeloma represents the second most common hematological malignancy.VELCADE is a small molecule to treat human malignancies. Its anti-neoplastic effect invovles several distinct mechanisms including inhibition of cell growth. Patients who have relapsed or are refractory to therapy, the standard of care is now VELCADE based on the results of previous clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent with the understanding that the consent may be w/d by the patient at any time w/o prejudice to future medical care.
2. Patient previously diagnosed with Multiple Myeloma (MM).
3. Patient previously tolerated 0.7, 1.0, or 1.3 mg/m2/dose of VELCADE alone or therapy combination and had at least a greater/equal 50% reduction in M-Protein upon completion of VELCADE therapy. The DOR prior to VELCADE greater/equal 4 months for the patient population.
4. It has been greater/equal 2 months since the patient's last VELCADE dose and the patient meets certain Lab criteria as per protocol.
5. Patient has a Karnosfsky performance status greater/equal 60%.
6. Patient has a life-expectancy greater than 3 months.
7. Patient has laboratory values (defined in protocol) within 14 days before enrollment.

Exclusion Criteria:

1. Patients with a Hx of PD, minimal response, or stable disease (SD)on first exposure to VELCADE.
2. Patient has received chemotherapy, radiotherapy, immunotherapy or experimental therapy to treat multiple myeloma since their last dose of VELCADE.
3. Patients who achieved a CR or PR but relapsed while on therapy.
4. Patient had major surgery w/in 2 wks before enrollment.
5. Patient has a Hx of allergic reaction to compounds containing boron or mannitol.
6. Patient has peripheral sensory neuropathy of Grade 2 w/pain or greater intensity.
7. Patient has cardiac amyloidosis.
8. Patient has poorly controlled hypertension, diabetes mellitus, or other serious medical or pysychiatric illness.
9. Patient is known to be human immunodeficiency virus (HIV)+.
10. Patient is known to be hepatitis B surface antigen-positive or has known active hepatitis C infection.
11. Patient has an active systemic infection requiring treatment.
12. Female patient is pregnant or breast-feeding. Confirmation must be established by a negative serum B-hCG.
13. Patient is currently enrolled in another clinical research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Walters, M.D., Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States